CLINICAL TRIAL: NCT00740545
Title: Essai thérapeutique randomisé Multicentrique en Double Insu, Comparant l'énoxaparine 40mg Versus Placebo, en Une Injection Sous-cutanée Quotidienne, Dans Les Fausses Couches spontanées récurrentes inexpliquées
Brief Title: Prevention of Unexplained Recurrent Abortion by Enoxaparine
Acronym: PREFIX
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped for futility
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RB06.050
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Alive and Viable Births
MeSH Terms: interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator)
  Interventions: Drug: placebo
- 1 (Experimental)
  Interventions: Drug: enoxaparine 40 mg daily

INTERVENTIONS:
Drug: enoxaparine 40 mg daily — Women inject ourselves every days with 40 mg of enoxaparine
  Arms: 1
Drug: placebo — Women inject ourselves every days with placebo
  Arms: 2

SUMMARY:
Standard investigations fail to reveal any apparent cause in 50% of the cases of recurrent spontaneous abortion. Prothrombotic mechanisms were initially evoked. Factor V Leiden, Prothrombin G20210A mutation and protein S deficiency are implicated in the meta-analysis of Rey (Lancet).However, they do not account for a large number of miscarriages.Gris JC and coworkers (Blood 2004)carried out an open trial, low-molecular-weight heparin versus low-dose aspirin, in women with one fetal loss and with a constitutional thrombophilic disorder. They conclude for a benefit action of Low-molecular-weight heparin. There is actually no trials concerning women with unexplained recurrent abortions and without known thrombophilia. Nevertheless,aspirin or enoxaparin are often prescribed. It is time to assess these practices. We therefore initiate a multisite, double blind randomized study, enoxaparine versus placebo, in women without known thrombophilia, which experienced unexplained recurrent abortions.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 45 years
* 2 or more consecutive spontaneous abortions before the 15th week of pregnancy
* Unexplained abortions
* No maternal or paternal characterized chromosomal aberration
* No Anti-phospholipid Syndrome
* No anatomical abnormality possibly responsible for abortion
* No Factor V Leiden
* No Prothrombin G20210A mutation
* No protein S deficiency
* No protein C deficiency
* No Anti thrombin 3 deficiency
* Proved pregnancy

Exclusion Criteria:

* Contraindications of enoxaparine 4000 U per day
* Women with risk of venous thromboembolism during pregnancy
* No regular anticoagulation or antiplatelet treatment
* Blood Hemoglobin level below 10g/dl
* Blood platelet level below 150 000/mm3
* Creatinine clearance below 30ml/mn
* Anomaly of the coagulation tests
* No informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 258 (Actual)
Dates: Start 2007-04; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Alive and Viable Births | number of born child healthy

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Pasquier, MD, Principal Investigator — Internal Medecine and pneumology department of university hospital of Brest (FRANCE)
Locations (7):
- France (7):
  - Centre Hospitalier Universitaire de Brest, Brest
  - Centre Hospitalier Régional Universitaire de Caen, Caen
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre Hospitalier Bretagne Sud, Lorient
  - Centre Hospitalier Nord Marseille, Marseille
  - Centre Hospitalier Universitaire de Rouen, Rouen
  - Centre Hospitalier Universitaire de St Etienne, Saint-Etienne

REFERENCES:
- [Derived] Pasquier E, de Saint Martin L, Bohec C, Chauleur C, Bretelle F, Marhic G, Le Gal G, Debarge V, Lecomte F, Denoual-Ziad C, Lejeune-Saada V, Douvier S, Heisert M, Mottier D. Enoxaparin for prevention of unexplained recurrent miscarriage: a multicenter randomized double-blind placebo-controlled trial. Blood. 2015 Apr 2;125(14):2200-5. doi: 10.1182/blood-2014-11-610857. Epub 2015 Jan 30. PMID 25636341